CLINICAL TRIAL: NCT02012205
Title: Safety and Efficacy of Wet Cupping on Persistent Non-specific Low Back Pain: A Randomized, Controlled, Open-label, Parallel-group
Brief Title: Wet Cupping in Non-specific Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Center for Complementary and Alternative Medicine, Saudi Arabia (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MOH044
Record Dates: First submitted 2013-12-03; First posted 2013-12-16 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: Persistent Non Specific Low Back Pain
Keywords: wet cupping - back pain - NSLBP - Saudi

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- wet cupping (Experimental): patient will receive wet cupping
  Interventions: Procedure: wet cupping
- control (No Intervention): not cupping

INTERVENTIONS:
Procedure: wet cupping — Participants assigned to the treatment group will receive wet-cupping therapy 3 times per week for 2 weeks
  Other Names: Hijamah
  Arms: wet cupping

SUMMARY:
Background: Persistent nonspecific low back pain (PNSLBP) is one of the most common low back pains worldwide. Many interventions were tried including wet cupping which is commonly used for pain conditions in Saudi Arabia and other parts in the world but without solid scientific evidence.

Aims: This study aims at determining safety and efficacy of wet cupping for treating PNSLBP.

Methods: This is a randomized wait-listed controlled clinical trial. Eligible patients with history of at least 3 months of PNSLBP will be randomized in to two groups, 45 patients each. The first group will be given wet-cupping treatment at two acupuncture points of urinary Bladder (BL) meridians among the BL23, BL24 and BL25, 6 times within 2 weeks. The second group will serve as a control group. Usual care, including providing brochures for exercise, general advice for PNSLBP and acetaminophen, will be allowed in both groups. Separate assessors participated in the outcome assessment. Investigators will use the 0 to100 numerical rating scale (NRS) for pain, the McGill Pain questionnaire for pain intensity (PPI) and the Oswestry Disability Questionnaire (ODQ), and to assess acetaminophen use and safety issues.

Expected Results: To provide data on the safety and effectiveness of wet cupping in treating PNSLBP and open the way for integrative medicine in Saudi Arabia

DETAILED DESCRIPTION:
Objectives:

To evaluate the effectiveness of wet cupping in the treatment of NSLBP:

1. Primary objective: To assess the effect of wet cupping on Pain (difference in the NRS from base to the end of two weeks) compared to the control group
2. Secondary objectives :

I-To compare Functioning (Oswestry Disability Questionnaire) from the base to the end of the two weeks of wet cupping sessions& two weeks later in the two groups II-To compare NRS from base to two weeks after the end of cupping III-To compare Number of Acetaminophen tables taken at the end of two weeks. IV-To evaluate Safety of wet cupping

SPECIFIC HYPOTHESIS: The hypothesis of this study is that the improvement of Numeric Rating Scale (NRS) for Pain at the end of the study will be greater in the Wet Cupping Treatment group than in the Control group

Overall Design: a randomised, waiting-list controlled, open-label, parallel trial.

* Study Type: Interventional
* Condition: Persistent Non Specific Low Back Pain (PNSLBP)

Case definition parameters:

* Low back pain: is defined as pain and discomfort, localized , below the costal margin and above the inferior gluteal folds, with or without referred leg pain.,
* Persistent low back pain: is defined as low back pain persisting for at least 12 weeks. We do not deal specifically with repeated, short bouts of pain.
* Nonspecific low back pain: is defined as" low back pain that is not attributable to a recognizable, known specific pathology (e.g. infection, tumour, osteoporosis, fracture, structural deformity, inflammatory disorder (e.g. ankylosing spondylitis), radicular syndrome or caudal equine syndrome)."

Study Design:

ELIGIBILITY:
Inclusion Criteria:

1. - Patients who have had non-specific low back pains at least 12 weeks now.
2. - Interested in using wet cupping therapy
3. - Age equal or more than 18 years up to 60 years of age.

Exclusion Criteria:

* 1-Patients who have low back pain due to specific and known etiological causes (infection, tumor, osteoporosis, ankylosing spondylitis, fracture, inflammatory process, radicular syndrome, cauda equinal syndrome).

  2-Patients who are inappropriate to the wet cupping treatment.
  * ◦AIDS, Active Hepatitis, Tuberculosis, Syphilis. (N.B.)Referring physicians will be advised to exclude patients with the above mentioned diseases.
  * ◦Patients who regularly take anticoagulants, antiplatelet drugs
  * ◦Anemia, thrombocytopenia
  * ◦Hemorrhagic disease like hemophilia
  * ◦Diabetes
  * ◦Severe cardiovascular disease
  * ◦Kidney diseases (renal failure, chronic renal disease)

    3-Patients who have experiences of wet cupping treatment during last 3 months. 4-Patients who have had treatment for low back pain during last 2 weeks. 5-Patients who are in pregnancy or have plan to conception. 6-Patients who have vertebra surgery or have plan of surgery.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2014-04; Primary Completion 2014-11 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
NRS | at the end of the two weeks wet cupping sessions.
  Difference in Numeric Rating Score at the base and at the end of two weeks of cupping sessions.

SECONDARY OUTCOMES:
Scores of the McGill Pain questionnaire for pain intensity (PPI) | at the end of two weeks of cupping sessions and two weeks later
  Change in the score from base line
the Oswestry Disability Questionnaire (ODQ), | at the end of two weeks of cupping sessions and two weeks later
  change in the score from the base line
Number of Participants with Serious and Non-Serious Adverse Events | at the last visit, one week after the end of the last sessions
  Differences in number of participants with Serious and Non-Serious Adverse Events.

CONTACTS AND LOCATIONS:
Overall Officials: Abdullah M AlBedah, MD, Principal Investigator — National Center for Complementary and Integrative Health (NCCIH); Mohamed K.M. Khalil, MD, Study Director — National Center for Complementary and Integrative Health (NCCIH)
Locations (3):
- Saudi Arabia (3):
  - King Fahad Specialist Hospital, Jeddah, Jeddah
  - King Fahad Hospital, Madinah, Madinah
  - Prince Salman Hospital, Riyadh, Riyadh Region

REFERENCES:
- [Derived] Al-Eidi SM, Mohamed AG, Abutalib RA, AlBedah AM, Khalil MKM. Wet Cupping-Traditional Hijamah Technique versus Asian Cupping Technique in Chronic Low Back Pain Patients: A Pilot Randomized Clinical Trial. J Acupunct Meridian Stud. 2019 Dec;12(6):173-181. doi: 10.1016/j.jams.2019.04.005. Epub 2019 Apr 24. PMID 31028971